CLINICAL TRIAL: NCT06963151
Title: Association of a HABIT-ILE Course and a Home Programme on the Bimanual Performance of Children Aged 3 to 5 Years With Cerebral Palsy: a Multicentre Randomised Controlled Trial of Non-inferiority
Brief Title: Association of a HABIT-ILE Course and a Home Programme on the Bimanual Performance of Children With Cerebral Palsy
Acronym: PARTNERSHIP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ildys (Other)
Collaborators: University Hospital, Angers (Other Government); LP3C, University of Rennes 2 (Unknown); Claude Bernard University (Other); IMT Atlantique Brest (Unknown); INSERM UMR 1101 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RI2023_001
Record Dates: First submitted 2025-03-17; First posted 2025-05-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy
Keywords: HABIT-ILE; Intensive motor therapy; Motor skill learning; Parental Coaching; Children; Additional Relavant MeSH Terms; Nervous System Diseases; Brain Damage, Chronic; Brain Diseases; Central Nervous System Diseases; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Nervous System Diseases; Brain Damage, Chronic; Brain Diseases; Central Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PARTNER (Experimental): Subjects will receive 35 hours of HABIT-ILE as camp format 3,5h/day, 5 days/week and 15 hours of home programme 1,5h/day, 5 day/week. These two procedures will be carried out concurrently over a 2-week period.
  Interventions: Other: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities
- HABIT-ILE (Experimental): Subjects will receive 50 hours of HABIT-ILE as camp format 5h/day, 5 days/week for two weeks.
  Interventions: Other: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities

INTERVENTIONS:
Other: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities — * Structured bimanual tasks training, with gradual increase in motor difficulty, requiring increased postural adjustments and the use of the lower extremities.
  * Home programme with parental coaching
  Arms: PARTNER
Other: Behavioral: Hand-Arm Bimanual Intensive Therapy Including Lower Extremities — - Structured bimanual tasks training, with gradual increase in motor difficulty, requiring increased postural adjustments and the use of the lower extremities.
  Arms: HABIT-ILE

SUMMARY:
This non-inferiority, mixed-methods, multicentre randomised controlled trial will compare the effects of functional changes and families' resources at 3 months of the PARTNER programme (35h HABIT-ILE + 15h home programme) with the reference HABIT-ILE programme (50h) on the bimanual performance (Assisting Hand Assessment [AHA]) of 66 children with unilateral CP aged 3 to 5 years.

DETAILED DESCRIPTION:
The PARTNERSHIP study will compare, for the first time, a mixed PARTNER camp modality, including a HABIT-ILE camp modality and a home programme modality, with parental coaching, to a reference HABIT-ILE modality.

The children in the PARTNER group will therefore spend 3.5 hours a day for 10 days in HABIT-ILE therapy, plus 1.5 hours a day for 10 days in home activities carried out by the family.

The children in the HABIT-ILE group will have 5 hours of HABIT-ILE therapy per day, the reference modality.

A non-inferiority, mixed-methods, multicentre randomised controlled trial will be conducted to compare the effectiveness of the PARTNER programme with the reference HABIT-ILE programme on the bimanual performance (Assisting Hand Assessment [AHA]) of children with unilateral CP aged 3 to 5 years. The secondary aims are to compare the 3-month effectiveness of the programmes on occupational performance, functional skills and upper limb activity levels, as well as families' resources, the parent-child relationship, the quantity and quality of resources available in the home to stimulate the child's motor development, and parental perceptions of their child's disability and their child's abilities (qualitative study). The tertiary aim is to conduct a cost-effectiveness analysis of care consumption in each group up to 6 months after the end of the programmes.

Target recruitment is 66 children (33 in each group) from 3 centres in France. Outcomes will be evaluated before the interventions, immediately after, at 3 months and up to 6 months for the cost-effectiveness analysis. Families in the PARTNER group will receive specific coaching and extensive support to perform the home programme. The coaching will focus on enhancing their resources.

ELIGIBILITY:
Inclusion Criteria:

1. Child with unilateral CP confirmed by a physician
2. Child aged between 3 years and 5 years 11 months (corrected age) at study entry
3. Ability to grasp a light object and lift it ≥15cm above the table using the affected hand.
4. Ability to understand instructions and complete all assessments.
5. Matched with another child based on age (± 3 months), CP aetiology, and Manual Ability Classification System (MACS) level.
6. Written informed consent obtained from a parent or legal guardian.
7. Commitment to having the same parent or guardian participate throughout the study.

Exclusion Criteria:

1. Diagnosis of ataxic CP.
2. Uncontrolled epilepsy.
3. History of botulinum toxin injection or surgery within 6 months of study entry or scheduled within 3 months of the intervention (ie, during the study period).
4. Visual or auditory deficits that could interfere with participation in the study.
5. Significant cognitive or behavioural disorder limiting the ability to follow instructions, as reported in discussions with the family, therapists and/or during a prior assessment

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Assisting Hand Assessment (AHA) | At the baseline (T0), at the end of the camp (T1: T0 + 21 + 2 days), and during the follow-up visit (T2: T0 + 90+2 days)
  The Assisting Hand Assessment (AHA) is a valid tool to assess children's ability to perform bimanual tasks, focusing on the functional use of the impaired hand. Its validity, reliability and responsiveness have been demonstrated, and it is regularly used in studies of children with unilateral CP.
  The raw AHA scores (min: 22 to max: 88) will be covered to a logit scale from 0 to 100 in order to obtain an interval scale, a proprety that the raw scores do not have. The conversion to this scale is based on a Rasch model. An increase in the AHA score indicates an improvement in the child's hability to perform bimanual taks.
  This study falls into the "Balanced Advantages" model of non-inferiority study designs. In this model, it is common to accept an inferiority level of 10 to 50% of the experimental treatment compared with the reference treatment. For this study, we set the accepted inferiority at -10% of the known values for the reference HABIT-ILE treatment; approximately 5 points.

SECONDARY OUTCOMES:
Canadian Measure of Occupational Performance (COPM) | At the baseline (T0), at the end of the camp (T1: T0+ 21+2 days), and during the follow-up visit (T2: T0+ 90+2 days)
  The Canadian Measure of Occupational Performance (COPM) will be used to define therapeutic goals, and to quantify the change in the child's performance and the parents' level of satisfaction for each functional goal. Using the COPM, the therapist conducts a semi-structured interview with the child's parent to identify difficulties in self-care, productivity, and leisure. The parent rates the importance of each indetified issue(1-10) and selects five priorities. For each, they rate their child's performance and their satisfaction with that performance (1-10, Higher ratings indicate greater importance, performance, and satisfaction). Average scores (out of 10) are calculated for performace and satisfaction. A change of two points or more is considered clinically significant.
  For this secondary outcome, the assumption is a maximum non-inferiority of 10% (T2-T0), ie, 0.4 points on average for the COPM, based on the results of Arenada et al..
Pediatric Evaluation of Disability Inventory Computer Adaptative Test (PEDI-CAT) | At the baseline (T0), at the end of the camp (T1: T0+ 21+2 days), and during the follow-up visit (T2: T0 +90+2 days)
  The Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT) will measure the change in functional skills in the domains of daily activities and mobility. These reliable questionnaires are used in clinical practice and research to determine changes in activity and participation in children with CP. These reliable questionnaires are used in clinical practice and research to determine changes in activity and participation in children with CP. The minimal score of PEDI CAT is 20 and the maximum 80, a higher score translates to higher function functional ability.
  For this secondary outcome, the assumption is a maximum non-inferiority of 10% (T2-T0), ie, 0.2 points for PEDI-CAT, based on the results of Arenada et al..
Gross motor activity and upper limb activity | 4 days at home before T0, during the camp, 4days at home before T2
  Gross motor activity (whole-body movements such as walking, cycling or jumping) and upper limb activity (movements of the arms, hands, and fingers, such as reaching, grasping or manipulating objects) will be measured using inertial sensors worn on each wrist and the trunk during the entire intervention time (35h+15h for the PARTNER group, 50h for the HABIT-ILE group). The main outcome will be the percentage of time spent performing movement during the sessions. The amount of activity performed at home out with sessions will also be measured in both groups.
Changes of family resources: World health organization quality of life - Bref (WHOQOL-Bref) | At the baseline (T0), at the end of the camp (T1: T0+ 21+2 days), and during the follow-up visit (T2: T0+ 90+2 days)
  To complete the questionnaire and participate in the semi-structured interviews, families will be asked to designate the child's main carer, who will agree to participate in the entire study and complete the questionnaires and interviews alone.
  The WHOQOL-Bref will measure parents' perceptions of their quality of life. This scale is derived from the WHOQOL-100 developed by the WHO (1995). It measures peopol's perception of their quality of life. The scale comprises 26 items divided into four areas: physical health, physiological health, social relationships end the environment. A hign score indicates a good quality of life, while a low score indicates a poorer quality of life. The 26 items are rated on a 5-point Likert scale (scores from 1 to 5). It is possible to obtain a score in each of the 4 domains (average score). These domain scores must be multiplied by 4 to be comparable with the WHOQOL-100. Two items can be analysed separately.
Changes of family resources: The Enabling Practice Scale (EPS) | At the baseline (T0), at the end of the camp (T1: T0+ 21+2 days), and during the follo-up visit (T2: T0+90+2 days)
  To complete the questionnaire and participate in the semi-structured interviews, families will be asked to designate the child's main carer, who will agree to participate in the entire study and complete the questionnaires and interviews alone.
  The Enabling Practice Scale (EPS) will be used to assess the parents' perception of the nature of the support provided by the referral workers. The total score will be analysed, EPS assesses parets' perceptions of the nature of the support provided by professionals providing care. This is a self-questionnaire containing 24 questions, each of which is scored on a 5-point Likert-type scale (from 1 to 5). The minimu score is 24, the maximum 120. A higher score indicates a higher level of enabling. The PES can be completed in 5 to 10 minutes. The overall score will be used in this study.
Changes of family resources: The Psychological Empowerment Scale (PES) | At the baseline (T0), at the end of the camp (T1: T0+ 21+2 days), and during the follow-up visit (T2: T0+ 90+2days)
  The Psychological Scale (PES) will be used to estimate changes in family empowerment in 3 dimensions: attitudes of control and competence, knowledge and kno-how, and participation behaviours. The Psychological Empowerment Scale (PES) evaluates parent's power to act on the basis of 32 items divided into three dimensions: attitudes of control and competence, knowledge and know-how, and participation behaviours. Each item is scored from 1 to 5 (minimum total score: 32, maximum: 160). A higher score indicates a higher level of empowerment. The total empowerment score will be analysed.
Changes of family resources: The Parental Stress Inventory (PSI) | At the baseline (T0), at the end of the camp (T1: T0+ 21±2 days)), and during the follow-up visit (T2: T0+ 90±2 days)
  The Parental Stress Inventory (PSI) will be used to measure the level of parental stress in the child's domain (eg, hyperactivity/distrac) ISP is a French translation of Abidin's Parental Stress Index (PSI). It measures the level of parental stress on the basis of 120 items belonging to two main categories: related to the child's domain: depression, feeling of competence, attachment, marital relationship, social isolation, parent's health, restrictions of the parent's role. The parent's answers are given on a likert-type scale ranging from 1 to 5, and it is possible to obtain a total stress score (raw score or percentage) or 15 sub-scores representing the child's and parent's domains. The inventory has been validated for use with parents of children with disabilities.
Home Environment for Motor Development Self-Report (AHEMD-SR) | At the baseline (T0), at the end of the camp (T1: T0+ 21±2 days)), and during the follow-up visit (T2: T0+ 90±2 days)
  The Affordances in the Home Environment for Motor Development Self-Report (AHEMD-SR) will be used to inventory the quantity and quality of resources available in the home to stimulate the child's motor development. The tool includes five dimensions: outdoor space, indoor space, variety of stimulation, gross motor toys, and fine motor toys. Each dimension is scored from 1 (very low) to 4 (very high), for a total score ranging from 5 to 20. Higher scores indicate a more favorable home environment for motor development.
Parent-Child Early Relational Assessment (PCERA) | At the baseline (T0), at the end of the camp (T1: T0+ 21±2 days), and during the follow-up visit (T2: T0+ 90±2 days)
  PCERA measures the quality of the relationship between a parent and child aged 1 to 4.5 years. PCERA includes a total of 65 individual items composed of 29 parental, 28 child, and 8 dyadic items. The PCERA manual outlines six subscales: (1) Parent Positive Affective Involvement, Sensitivity, and Responsiveness; (2) Parent Negative Affect and Behavior; (3) Infant Positive Affect, Communication, and Social Skills; (4) Infant Dysregulation and Irritability; (5) Dyadic Mutuality and Reciprocity; and (6) Dyadic Tension. All items are coded into a three-point scale describing areas of concern (scores 1 and 2), areas of some concern (score 3) and areas of strength (scores 4 and 5). The overall minimum score is 65 and the maximal 325. Higher PCERA scores reflect more positive affect and/or behavior (subscales 1, 3 and 5). Consequently, higher scores on subscales 2, 4, and 6 indicate lower levels of negative affect and/or behavior.
Parental representations: PARTNER programme | At the baseline (T0), and during the follow-up visit (T2: T0+ 90±2 days)
  The impact of the PARTNER programme on parental representations of their child's disability and abilities will be assessed using semi-structured interviews. Changes in the parents' representations from before to after the programme will be assessed, and representations will be compared between each group with a sample of parents. The quality of responses will be related to the scores obtained on the various quantitative measures.
Cost-effectiveness analysis | From baseline (T0) to the end of the camp (T1: T0+ 21±2 days
  The costs (structural and family) will be measured for children taking part in both types of camp The cost-effectiveness analysis will be conducted by calculating the incremental cost-effectiveness ratio (ICER), defined as the ratio between the average difference in costs between the intervention and the comparator (ΔC) and the average difference in effectiveness measured by the improvement in the AHA score (ΔE). The uncertainty around the ICER will be explored using a cost-effectiveness plane, and a cost-effectiveness acceptability curve (CEAC) will estimate the probability that the intervention is cost-effective for different willingness-to-pay (WTP) thresholds. Non-parametric tests (Mann-Whitney (Wilcoxon) test for two groups) will be implemented for cost comparison.
Impact on care consumption | From baseline (T0) to 6 months post intervention.
  The actual care consumption of each child will be collected automatically by consulting the RNIPP register (National Register of Identification of Natural Persons).
  - The difference in care consumption between groups up to 6 months after the end of the intervention will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe BAILLY, Principal Investigator — Fondation Ildys
Locations (1):
- Fondation ILDYS, Brest, France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tedla JS, Asiri F, Reddy RS, Gular K, Kakaraparthi VN, Sangadala DR, Dixit S, Alamri AM, Narne VK, Alasmari RAM, Dhafer OA, Al Shamer MA. Caregiver's Quality of Life Among Children with Cerebral Palsy in the Kingdom of Saudi Arabia, and Various Influencing Factors: A Single Cohort Study. J Multidiscip Healthc. 2023 Nov 29;16:3705-3714. doi: 10.2147/JMDH.S440190. eCollection 2023. Erratum In: J Multidiscip Healthc. 2023 Dec 23;16:4211-4212. doi: 10.2147/JMDH.S456266. PMID 38050486
- [Background] Laister D, Vivanti G, Marschik PB, Fellinger J, Holzinger D. Enhancement of Social Communication Behaviors in Young Children With Autism Affects Maternal Stress. Front Psychiatry. 2021 Dec 7;12:797148. doi: 10.3389/fpsyt.2021.797148. eCollection 2021. PMID 34950076
- [Background] Krumlinde-Sundholm L, Holmefur M, Kottorp A, Eliasson AC. The Assisting Hand Assessment: current evidence of validity, reliability, and responsiveness to change. Dev Med Child Neurol. 2007 Apr;49(4):259-64. doi: 10.1111/j.1469-8749.2007.00259.x. PMID 17376135
- [Background] Karstad SB, Bjorseth A, Lindstedt J, Brenne AS, Steihaug H, Elvrum AG. Parental Coping, Representations, and Interactions with Their Infants at High Risk of Cerebral Palsy. J Clin Med. 2022 Dec 29;12(1):277. doi: 10.3390/jcm12010277. PMID 36615077
- [Background] Kang M, Smith E, Goldsmith CH, Switzer L, Rosenbaum P, Wright FV, Fehlings D. Documenting change with the Canadian Occupational Performance Measure for children with cerebral palsy. Dev Med Child Neurol. 2020 Oct;62(10):1154-1160. doi: 10.1111/dmcn.14569. Epub 2020 Jun 3. PMID 32491226
- [Background] Holmefur M, Aarts P, Hoare B, Krumlinde-Sundholm L. Test-retest and alternate forms reliability of the assisting hand assessment. J Rehabil Med. 2009 Nov;41(11):886-91. doi: 10.2340/16501977-0448. PMID 19841839
- [Background] Bonden H, Jahnsen RB, Klevberg GL. Self-care and hand function in preschool children with unilateral or bilateral cerebral palsy: A cross-sectional study. Child Care Health Dev. 2024 Jan;50(1):e13208. doi: 10.1111/cch.13208. Epub 2023 Dec 11. PMID 38083836
- [Background] Araneda R, Ebner-Karestinos D, Paradis J, Klocker A, Saussez G, Demas J, Bailly R, Bouvier S, Carton de Tournai A, Herman E, Souki A, Le Gal G, Nowak E, Sizonenko SV, Newman CJ, Dinomais M, Riquelme I, Guzzetta A, Brochard S, Bleyenheuft Y. Changes Induced by Early Hand-Arm Bimanual Intensive Therapy Including Lower Extremities in Young Children With Unilateral Cerebral Palsy: A Randomized Clinical Trial. JAMA Pediatr. 2024 Jan 1;178(1):19-28. doi: 10.1001/jamapediatrics.2023.4809. PMID 37930692
- [Derived] Demas J, Jacquemot D, Bouvier S, Goff ML, Carcreff L, Dinomais M, Vuillerot C, Brochard S, Dubois A, Bailly R. Is PARTNER, a hybrid HABIT-ILE programme with parent coaching, as effective as standard HABIT-ILE in children with cerebral palsy aged 3-5? A protocol for a multicentre, randomised controlled trial. BMJ Open. 2025 Sep 16;15(9):e105076. doi: 10.1136/bmjopen-2025-105076. PMID 40962347